CLINICAL TRIAL: NCT00586651
Title: An Open-Label Study of Oral CEP-701 in Patients With Polycythemia Vera or Essential Thrombocytosis With the JAK2 V617F Mutation
Brief Title: Open-Label Study of Oral CEP-701 (Lestaurtinib) in Patients With Polycythemia Vera or Essential Thrombocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0701/2030/ON/US
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Polycythemia Vera; Essential Thrombocytosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — lestaurtinib

ARMS (1):
- lestaurtinib (Experimental)
  Interventions: Drug: lestaurtinib

INTERVENTIONS:
Drug: lestaurtinib — 60 mg bid - 120 mg bid for an 18 weeks (126 days) treatment duration

SUMMARY:
This is an 18-week open-label, multicenter study to evaluate the efficacy and tolerability of CEP-701 (lestaurtinib) treatment in patients with Polycythemia Vera (PV) and patients with Essential Thrombocytosis (ET).

DETAILED DESCRIPTION:
This is an 18-week open-label, multicenter study to evaluate the efficacy and tolerability of CEP-701 (lestaurtinib) treatment at a dosage of 80 mg bid for 18 weeks (126 days) in patients with Polycythemia Vera (PV) who have abnormal baseline neutrophil counts or require hydroxyurea therapy and patients with Essential Thrombocytosis (ET) who require hydroxyurea therapy for disease control.

ELIGIBILITY:
Inclusion Criteria:

* The patient has polycythemia vera (PV) or essential thrombocytosis (ET).
* The patient has a detectable JAK2 V617F mutation.
* Patients with PV have at least 1 of the following risk factors:

  1. neutrophil count greater than 7000/mm3
  2. receiving hydroxyurea treatment
* Patients with ET are receiving concomitant hydroxyurea.
* The patient has an ECOG performance score of 0, 1, or 2.

Exclusion Criteria:

* The patient has bilirubin levels or aspartate transaminases (AST) levels within exclusionary ranges.
* patient has serum creatinine concentrations within exclusionary ranges.
* patient has an untreated or progressive infection.
* patient has any physical or psychiatric condition that may compromise participation in the study.
* has a history of venous or arterial thrombosis within 6 months.
* use of hydroxyurea has been initiated or escalated in the month prior to screening.
* has active gastrointestinal ulceration or bleeding.
* patient has used an investigational drug within the past 30 days.
* patient is being treated with anagrelide.
* patient has previously taken CEP-701 (lestaurtinib).
* patient has hypersensitivity to CEP-701 (lestaurtinib) or any component of CEP-701 (lestaurtinib).
* patient has received interferon within the past 30 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine whether a specific reduction in the JAK2 V617F allele has been indicated in this study. | 18 weeks +

SECONDARY OUTCOMES:
- improvements in hemoglobin values, neutrophil count, and platelet count. - reduction in dose of hydroxyurea - reduction in splenic enlargement - rate of phlebotomy | 18 weeks +

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - NY Presbyterian-Cornell, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Hexner E, Roboz G, Hoffman R, Luger S, Mascarenhas J, Carroll M, Clementi R, Bensen-Kennedy D, Moliterno A. Open-label study of oral CEP-701 (lestaurtinib) in patients with polycythaemia vera or essential thrombocythaemia with JAK2-V617F mutation. Br J Haematol. 2014 Jan;164(1):83-93. doi: 10.1111/bjh.12607. Epub 2013 Oct 28. PMID 24903629